CLINICAL TRIAL: NCT00354549
Title: Bevacizumab and Erlotinib First-Line Therapy in Advanced Non-Squamous Non-Small-Cell Lung Cancer (Stage IIIB/IV) Followed by Platinum-Based Chemotherapy at Disease Progression. A Multicenter Phase II Trial
Brief Title: Bevacizumab and Erlotinib Followed by Cisplatin or Carboplatin and Gemcitabine in Treating Patients With Newly Diagnosed or Recurrent Stage IIIB or Stage IV NSCLC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Swiss Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SAKK 19/05; EU-20614
Record Dates: First submitted 2006-07-19; First posted 2006-07-20 (Estimated); Last update posted 2019-05-15 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; bronchoalveolar cell lung cancer; large cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Bevacizumab; Erlotinib Hydrochloride; Gemcitabine; Cisplatin; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: bevacizumab + erlotinib hydrochloride — Patients receive bevacizumab IV over 90 minutes on day 1 and oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.
Drug: gemcitabine hydrochloride + cisplatin or carboplatin — Beginning within 3 weeks of documented disease progression, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. They also receive cisplatin IV over 1 hour or carboplatin IV over 30 minutes on day 1. Treatment with gemcitabine hydrochloride with either cisplatin or carboplatin repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

SUMMARY:
RATIONALE: Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, carboplatin, and gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving bevacizumab together with erlotinib followed by cisplatin or carboplatin and gemcitabine at disease progression may be an effective treatment for non-small cell lung cancer.

PURPOSE: This phase II trial is studying how well giving bevacizumab together with erlotinib followed by cisplatin or carboplatin and gemcitabine works in treating patients with newly diagnosed or recurrent stage IIIB or stage IV non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the efficacy of bevacizumab and erlotinib hydrochloride as initial therapy in patients with newly diagnosed or recurrent stage IIIB or IV non-squamous non-small cell lung cancer (NSCLC).

Secondary

* Assess the safety of bevacizumab and erlotinib hydrochloride as initial therapy in these patients.
* Assess the quality of life (QOL) in patients treated with bevacizumab and erlotinib hydrochloride.
* Assess the efficacy and safety of subsequent cisplatin or carboplatin in combination with gemcitabine hydrochloride in patients who have disease progression.
* Assess the QOL in patients treated with subsequent cisplatin or carboplatin in combination with gemcitabine hydrochloride at disease progression.

Tertiary

* Identify novel biomarkers in predicting response to therapy and toxicity in patients treated with bevacizumab and erlotinib hydrochloride as initial therapy.

OUTLINE: This is a multicenter, prospective, open-label study.

Patients receive bevacizumab IV over 90 minutes on day 1 and oral erlotinib hydrochloride once daily on days 1-21. Treatment repeats every 3 weeks in the absence of disease progression or unacceptable toxicity.

Beginning within 3 weeks of documented disease progression, patients receive gemcitabine hydrochloride IV over 30 minutes on days 1 and 8. They also receive cisplatin IV over 1 hour or carboplatin IV over 30 minutes on day 1. Treatment with gemcitabine hydrochloride with either cisplatin or carboplatin repeats every 21 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

Quality of life is assessed at baseline and periodically during study treatment.

After completion of study treatment, patients are followed every 3 months.

PROJECTED ACCRUAL: A total of 101 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-squamous non-small cell lung cancer (NSCLC)

  * Newly diagnosed or recurrent disease
* Meets 1 of the following staging criteria:

  * Stage IIIB disease, meeting both of the following criteria:

    * Proven malignant effusion or supraclavicular node involvement (i.e., N3 supraclavicular nodes)
    * Not a candidate for curative multimodality treatment or surgery
  * Stage IV disease
* Measurable disease, defined as ≥ 1 lesion (outside of irradiated areas) that can be measured in ≥ 1 dimension as ≥ 10 mm by spiral or multi-slice CT scan or MRI
* Immediate chemotherapy not clinically mandatory in the judgement of the investigator
* No intrathoracic large, centrally located tumors and/or cavitary lesions invading or abutting major blood vessels
* No evidence of clinically active interstitial lung disease

  * Patients with chronic stable radiographic changes who are asymptomatic are eligible
* No small cell lung cancer (SCLC), squamous NSCLC, or combined SCLC-NSCLC tumors
* No brain metastases

PATIENT CHARACTERISTICS:

* WHO performance status 0-1
* Hemoglobin ≥ 10 g/dL
* Absolute neutrophil count ≥ 1,500/mm³
* Thrombocyte count ≥ 100,000/mm³
* Bilirubin ≤ 1.5 times upper limit of normal (ULN)
* ALT ≤ 2.5 times ULN (5 times ULN if liver metastases present)
* Alkaline phosphatase ≤ 2.5 times ULN (5 times ULN if bone metastases present)
* Quick ≥ 70% OR INR ≤ 1.5
* Creatinine ≤ 2.0 times ULN
* Proteinuria ≤ 2+ by urine dipstick
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 12 months after completion of study treatment
* Able to understand trial information given by the investigator and complete quality of life questionnaire
* No pre-existing condition that would preclude swallowing and/or absorption of oral medication
* No prior or concurrent malignancies, except for the following:

  * Malignancy for which the minimum relapse-free interval is ≥ 5 years
  * Nonmelanoma skin cancer or adequately treated carcinoma in situ of the cervix
* No other medical condition that would preclude study participation, including any of the following:

  * Unstable or uncompensated respiratory, cardiac, hepatic, or renal disease
  * Active infection
  * Uncontrolled diabetes mellitus
  * Hypertension ≥ 150/100 mm Hg despite treatment
  * Myocardial infarction within the past 3 months
  * History of hemorrhagic disorders
  * Non-healing wound, ulcer, or bone fracture
* No clinical history of coagulopathy or thrombosis
* No hemoptysis or hematemesis ≥ grade 2 (defined as bright red blood of ≥ 5 mL per episode) within the past 6 months
* No known hypersensitivity to study drug(s) or to any other component of the study drugs
* No significant traumatic injury within the past 28 days
* No serious underlying medical condition that would impair the ability of the patient to participate in the trial or that would preclude use of study drugs
* No cerebrovascular accident or other CNS bleeding within the past 6 months

PRIOR CONCURRENT THERAPY:

* At least 4 weeks since prior radiotherapy and recovered

  * No prior radiotherapy to lesion(s) selected for measurement
* No prior chemotherapy for advanced disease

  * At least 6 months since prior neoadjuvant or adjuvant systemic chemotherapy for NSCLC
  * Prior intrapleural or intrapericardial local chemotherapy allowed
* No prior endothelial growth factor and/or vascular endothelial growth factor (receptor)-targeted therapy for NSCLC
* More than 28 days since prior major surgical procedure or open biopsy
* More than 30 days since prior treatment in another clinical trial
* No concurrent anticoagulants (e.g., phenprocoumon, acenocoumarol, or full-dose warfarin or heparin)
* No concurrent full-dose continuous use of non-steroid anti-inflammatory drugs (NSAIDs)
* No concurrent aspirin or clopidogrel bisulfate

  * Low-dose aspirin (≤ 325 mg daily) may be continued in patients at high risk for arterial thromboembolic disease
* No other concurrent drugs contraindicated for use with the study drugs, according to the Swissmedic-approved product information
* No other concurrent experimental drugs or anticancer therapy, including chemotherapy, immunotherapy, or hormone therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2006-01; Primary Completion 2009-04 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Disease stabilization (DS) (complete response [CR], partial response [PR], or stable disease [SD]) as assessed by RECIST criteria after 12 weeks of treatment with bevacizumab and erlotinib hydrochloride | 12 weeks

SECONDARY OUTCOMES:
DS as assessed by RECIST criteria after 6 and 18 weeks of treatment with bevacizumab and erlotinib hydrochloride | 6 and 18 weeks
Objective response (CR or PR) as assessed by RECIST criteria after 6, 12, and 18 weeks of treatment with bevacizumab and erlotinib hydrochloride | 6, 12 and 18 weeks
Best overall response when treated with bevacizumab and erlotinib hydrochloride | Until treatment ends
Adverse events (AEs) when treated with bevacizumab and erlotinib hydrochloride | Until treatment ends
Time to progression (TTP) when treated with bevacizumab and erlotinib hydrochloride | Until treatment ends
Time to treatment failure (TTF) when treated with bevacizumab and erlotinib hydrochloride | Until treatment ends
Quality of life (QOL) when treated with bevacizumab and erlotinib hydrochloride | Until treatment ends
Objective response (CR or PR) when treated with chemotherapy | Until treatment ends
Unexpected adverse drug reaction | Until treatment ends
QOL when treated with chemotherapy | Periodically
Overall survival (OS) in patients treated with bevacizumab and erlotinib hydrochloride and in patients treated with subsequent chemotherapy at disease progression | life-long

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Zappa, MD, Study Chair — Istituto Oncologico della Svizzera Italiana - Ospedale San Giovanni
Locations (2):
- Switzerland (2):
  - Universitaetsspital-Basel, Basel
  - Oncology Institute of Southern Switzerland, Bellinzona

REFERENCES:
- [Result] Zappa F, Droege C, Betticher D, von Moos R, Bubendorf L, Ochsenbein A, Gautschi O, Oppliger Leibundgut E, Froesch P, Stahel R, Hess T, Rauch D, Schmid P, Mayer M, Crowe S, Brauchli P, Ribi K, Pless M; Swiss Group for Clinical Cancer Research (SAKK). Bevacizumab and erlotinib (BE) first-line therapy in advanced non-squamous non-small-cell lung cancer (NSCLC) (stage IIIB/IV) followed by platinum-based chemotherapy (CT) at disease progression: a multicenter phase II trial (SAKK 19/05). Lung Cancer. 2012 Dec;78(3):239-44. doi: 10.1016/j.lungcan.2012.08.017. Epub 2012 Sep 23. PMID 23009726
- [Result] Baty F, Joerger M, Fruh M, Klingbiel D, Zappa F, Brutsche M. 24h-gene variation effect of combined bevacizumab/erlotinib in advanced non-squamous non-small cell lung cancer using exon array blood profiling. J Transl Med. 2017 Mar 30;15(1):66. doi: 10.1186/s12967-017-1174-z. PMID 28359318
- [Result] Franzini A, Baty F, Macovei II, Durr O, Droege C, Betticher D, Grigoriu BD, Klingbiel D, Zappa F, Brutsche MH. Gene Expression Signatures Predictive of Bevacizumab/Erlotinib Therapeutic Benefit in Advanced Nonsquamous Non-Small Cell Lung Cancer Patients (SAKK 19/05 trial). Clin Cancer Res. 2015 Dec 1;21(23):5253-63. doi: 10.1158/1078-0432.CCR-14-3135. Epub 2015 Apr 28. PMID 25922429
- [Result] Joerger M, Baty F, Fruh M, Droege C, Stahel RA, Betticher DC, von Moos R, Ochsenbein A, Pless M, Gautschi O, Rothschild S, Brauchli P, Klingbiel D, Zappa F, Brutsche M. Circulating microRNA profiling in patients with advanced non-squamous NSCLC receiving bevacizumab/erlotinib followed by platinum-based chemotherapy at progression (SAKK 19/05). Lung Cancer. 2014 Aug;85(2):306-13. doi: 10.1016/j.lungcan.2014.04.014. Epub 2014 May 29. PMID 24928469